CLINICAL TRIAL: NCT00658619
Title: Safety and Efficacy of Brimonidine Intravitreal Implant in Patients With Geographic Atrophy Due to AMD
Brief Title: Safety and Efficacy of Brimonidine Intravitreal Implant in Patients With Geographic Atrophy Due to Age-related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 190342-032D
Record Dates: First submitted 2008-04-11; First posted 2008-04-15 (Estimated); Results first posted 2013-04-26 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Brimonidine Tartrate; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 400 µg Brimonidine Tartrate Implant Stage 1 (Other): Stage 1: 400 µg brimonidine tartrate implant in the study eye and sham in the fellow eye on Day 1 and Month 6.
  Interventions: Drug: 400 µg Brimonidine Tartrate Implant; Other: Sham (no implant)
- 200 µg Brimonidine Tartrate Implant Stage 1 (Other): Stage 1: 200 µg brimonidine tartrate implant in the study eye and sham in the fellow eye on Day 1 and Month 6.
  Interventions: Drug: 200 µg Brimonidine Tartrate Implant; Other: Sham (no implant)
- 400 µg Brimonidine Tartrate Implant Stage 2 (Other): Stage 2: 400 µg brimonidine tartrate implant in the study eye and sham in the fellow eye on Day 1 and Month 6.
  Interventions: Drug: 400 µg Brimonidine Tartrate Implant; Other: Sham (no implant)
- 200 µg Brimonidine Tartrate Implant Stage 2 (Other): Stage 2: 200 µg brimonidine tartrate implant in the study eye and sham in the fellow eye on Day 1 and Month 6.
  Interventions: Drug: 200 µg Brimonidine Tartrate Implant; Other: Sham (no implant)
- Sham (no implant) Stage 2 (Sham Comparator): Stage 2: sham in both eyes on Day 1 and Month 6.
  Interventions: Other: Sham (no implant)

INTERVENTIONS:
Drug: 400 µg Brimonidine Tartrate Implant — 400 µg brimonidine tartrate implant in the study eye on Day 1 and Month 6.
  Other Names: Brimonidine Tartrate PS DDS®
  Arms: 400 µg Brimonidine Tartrate Implant Stage 1; 400 µg Brimonidine Tartrate Implant Stage 2
Drug: 200 µg Brimonidine Tartrate Implant — 200 µg brimonidine tartrate implant in the study eye on Day 1 and Month 6.
  Other Names: Brimonidine Tartrate PS DDS®
  Arms: 200 µg Brimonidine Tartrate Implant Stage 1; 200 µg Brimonidine Tartrate Implant Stage 2
Other: Sham (no implant) — Sham in one or both eyes on Day 1 and Month 6.

SUMMARY:
Stage 1 is a patient-masked, dose-escalation, safety evaluation of brimonidine intravitreal implant. Patients will receive implant in one eye and "sham" treatment (meaning no treatment) in the fellow eye. Stage 2 will begin after 1 month of safety has been evaluated for Stage 1. Stage 2 is a randomized, double-masked, dose-response, sham-controlled evaluation of the safety and efficacy of brimonidine intravitreal implant in patients with geographic atrophy from age-related macular degeneration. Patients will be followed for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Geographic atrophy in both eyes due to age-related macular degeneration
* Visual acuity between 20/40 to 20/320

Exclusion Criteria:

* Known allergy to brimonidine
* Uncontrolled systemic disease or infection of the eye
* Recent eye surgery or injections in the eye
* Female patients who are pregnant, nursing or planning a pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2008-05-01 (Actual); Primary Completion 2010-06-01 (Actual); Study Completion 2011-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (7):
- Abilene, Texas, United States
- Sydney, New South Wales, Australia
- Karlsruhe, Germany
- Udine, Italy
- Makati City, Philippines
- Coimbra, Portugal
- Seoul, South Korea

REFERENCES:
- [Derived] Kuppermann BD, Patel SS, Boyer DS, Augustin AJ, Freeman WR, Kerr KJ, Guo Q, Schneider S, Lopez FJ; Brimo DDS Gen 1 Study Group. PHASE 2 STUDY OF THE SAFETY AND EFFICACY OF BRIMONIDINE DRUG DELIVERY SYSTEM (BRIMO DDS) GENERATION 1 IN PATIENTS WITH GEOGRAPHIC ATROPHY SECONDARY TO AGE-RELATED MACULAR DEGENERATION. Retina. 2021 Jan 1;41(1):144-155. doi: 10.1097/IAE.0000000000002789. PMID 32134802

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Stage 1 of the study was a patient-masked, dose-escalation, paired-eye comparison and the Investigator was not masked. Stage 2 was a parallel-group, sham-controlled, paired-eye comparison. Investigators were masked as to dose received for patients in the active treatment groups. No patients from Stage 1 were enrolled in Stage 2.
Period: Overall Study
Arm/Group | 400 µg Brimonidine Tartrate Implant Stage 1 | 200 µg Brimonidine Tartrate Implant Stage 1 | 400 µg Brimonidine Tartrate Implant Stage 2 | 200 µg Brimonidine Tartrate Implant Stage 2 | Sham (no Implant) Stage 2
Started | 3 | 3 | 41 | 49 | 23
Completed | 3 | 2 | 31 | 37 | 21
Not Completed | 0 | 1 | 10 | 12 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 400 µg Brimonidine Tartrate Implant Stage 1 | 200 µg Brimonidine Tartrate Implant Stage 1 | 400 µg Brimonidine Tartrate Implant Stage 2 | 200 µg Brimonidine Tartrate Implant Stage 2 | Sham (no Implant) Stage 2 | Total
Number analyzed (Participants) | 3 | 3 | 41 | 49 | 23 | 119
Age, Continuous [Mean (Standard Deviation); unit: Years] | 85.0 (3.61) | 79.0 (3.00) | 75.6 (8.78) | 77.0 (9.13) | 78.4 (5.80) | 77.0 (8.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 27 | 28 | 12 | 72
  Male | 0 | 1 | 14 | 21 | 11 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Size of Geographic Atrophy Lesion Area in the Study Eye
Description: Change from baseline in size of geographic atrophy lesion area in the study eye is based on fundus photography as read by an independent Reading Center. Photographs are taken with a specialized microscope with an attached camera to photograph the interior of the eye, including the retina and optic disc. A positive change from baseline indicates an increase in size of geographic atrophy lesion area (worsening; disease progression). Data are reported in disc area where 1 disc area = 1.767 millimeters squared (mm^2).
Time Frame: Baseline, Month 12
Population: Intent-to-Treat: All randomized patients who participated in Stage 2
Measure: Mean (Standard Deviation); unit: Disc Area
Arm/Group | 400 µg Brimonidine Tartrate Implant Stage 2 | 200 µg Brimonidine Tartrate Implant Stage 2 | Sham (no Implant) Stage 2
Number analyzed (Participants) | 41 | 49 | 23
Disc Area
  Baseline | 6.219 (3.9524) | 6.897 (4.6397) | 5.526 (4.7890)
  Change from Baseline at Month 12 | 0.898 (0.7520) | 1.006 (0.7858) | 1.239 (1.1645)

2. Secondary Outcome: Change From Baseline in Size of Geographic Atrophy Lesion Area in the Study Eye
Description: as for outcome 1
Time Frame: Baseline, Month 3, Month 6, Month 9, Month 18, Month 24
Population: Intent-to-Treat: All randomized patients who participated in Stage 2
Measure: Mean (Standard Deviation); unit: Disc Area
Groups:
- 200 µg Brimonidine Tartrate Implant Stage 2: Stage 2: 200 µg brimonidine tartrate implant in study eye and sham in fellow eye on Day 1 and Month 6.
Arm/Group | 400 µg Brimonidine Tartrate Implant Stage 2 | 200 µg Brimonidine Tartrate Implant Stage 2 | Sham (no Implant) Stage 2
Number analyzed (Participants) | 41 | 49 | 23
Disc Area
  Baseline | 6.219 (3.9524) | 6.897 (4.6397) | 5.526 (4.7890)
  Change from Baseline at Month 3 | 0.182 (0.3353) | 0.117 (0.6612) | 0.399 (0.3713)
  Change from Baseline at Month 6 | 0.482 (0.6325) | 0.570 (0.5749) | 0.609 (0.5474)
  Change from Baseline at Month 9 | 0.641 (0.6847) | 0.798 (0.6424) | 0.857 (0.7267)
  Change from Baseline at Month 18 | 1.306 (1.0164) | 1.413 (1.0291) | 1.697 (1.4185)
  Change from Baseline at Month 24 | 1.744 (1.4010) | 1.991 (1.4469) | 2.178 (1.7042)

3. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening.
Time Frame: Baseline, 24 Months
Population: Intent-to-Treat: All randomized patients who participated in Stage 2
Measure: Mean (Standard Deviation); unit: Number of Letters Read Correctly
Arm/Group | 400 µg Brimonidine Tartrate Implant Stage 2 | 200 µg Brimonidine Tartrate Implant Stage 2 | Sham (no Implant) Stage 2
Number analyzed (Participants) | 41 | 49 | 23
Number of Letters Read Correctly
  Baseline | 54.8 (12.89) | 52.1 (13.91) | 53.7 (10.71)
  Change from Baseline at 24 Months | -5.0 (13.77) | -3.2 (12.87) | -3.3 (12.98)

4. Secondary Outcome: Change From Baseline in Contrast Sensitivity in the Study Eye
Description: Change from baseline in contrast sensitivity in the study eye is measured using a Pelli-Robson contrast sensitivity chart at 1 meter. The contrast sensitivity chart contains letters that are darkest at the top and then get progressively lighter. Scores range from 0 to 48 and are based on the number of letters read correctly. A negative change from baseline indicates a worsening in contrast sensitivity and a positive change from baseline indicates an improvement.
Time Frame: Baseline, 24 Months
Population: Intent-to-Treat: All randomized patients who participated in Stage 2
Measure: Mean (Standard Deviation); unit: Number of Letters Read Correctly
Arm/Group | 400 µg Brimonidine Tartrate Implant Stage 2 | 200 µg Brimonidine Tartrate Implant Stage 2 | Sham (no Implant) Stage 2
Number analyzed (Participants) | 41 | 49 | 23
Number of Letters Read Correctly
  Baseline | 23.7 (5.60) | 22.1 (5.76) | 21.7 (7.56)
  Change from Baseline at 24 Months | -0.9 (4.33) | 1.1 (7.22) | 0.6 (7.49)

5. Secondary Outcome: Change From Baseline in Reading Speed in the Study Eye
Description: Change from baseline in reading speed in the study eye is assessed using modified Bailey-Lovie word charts. Patients read the chart for 2 minutes and the numbers of words read correctly per minute are totaled. An increase in the number of words read correctly indicates an improvement and a decrease in the number of words read correctly indicates a worsening.
Time Frame: Baseline, 24 Months
Population: Intent-to-Treat: All randomized patients who participated in Stage 2
Measure: Mean (Standard Deviation); unit: Words per Minute (wpm)
Arm/Group | 400 µg Brimonidine Tartrate Implant Stage 2 | 200 µg Brimonidine Tartrate Implant Stage 2 | Sham (no Implant) Stage 2
Number analyzed (Participants) | 41 | 49 | 23
Words per Minute (wpm)
  Baseline | 10.21 (8.532) | 9.62 (9.224) | 8.72 (6.832)
  Change from Baseline at 24 Months | -1.15 (5.527) | -0.28 (7.035) | 0.45 (4.705)

ADVERSE EVENTS:
Description: The Safety Population was used for adverse events (AEs) and serious adverse events (SAEs) and included all patients who were enrolled and treated in the study. For Ocular AEs, only those occurring in the study eye are reported in the "Other Adverse Events" section. For SAEs, all ocular events are reported, regardless of eye.
Groups:
- 400 µg Brimonidine Tartrate Implant: Stage 1 and 2 combined: 400 µg brimonidine tartrate implant in the study eye and sham in the fellow eye on Day 1 and Month 6.
- 200 µg Brimonidine Tartrate Implant: Stage 1 and 2 combined: 200 µg brimonidine tartrate implant in the study eye and sham in the fellow eye on Day 1 and Month 6.
Arm/Group | 400 µg Brimonidine Tartrate Implant | 200 µg Brimonidine Tartrate Implant | Sham (no Implant) Stage 2
Serious Adverse Events (participants affected / at risk) | 14/43 | 20/51 | 9/23
Other Adverse Events (participants affected / at risk) | 38/43 | 47/51 | 20/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 400 µg Brimonidine Tartrate Implant (N=43) | 200 µg Brimonidine Tartrate Implant (N=51) | Sham (no Implant) Stage 2 (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Angina Unstable (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 2 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0
Aortic Valve Stenosis (Cardiac disorders) | 0 | 1 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1 | 0
Mitral Valve Stenosis (Cardiac disorders) | 0 | 1 | 0
Sick Sinus Syndrome (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Visual Acuity Reduced (Eye disorders) | 1 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal Stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea Infectious (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung Squamous Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 2 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Intracranial Aneurysm (Nervous system disorders) | 0 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0 | 0
Stress Urinary Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0
Pulmonary Vascular Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Aortic Stenosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 400 µg Brimonidine Tartrate Implant (N=43) | 200 µg Brimonidine Tartrate Implant (N=51) | Sham (no Implant) Stage 2 (N=23)
Anaemia (Blood and lymphatic system disorders) | 1 | 5 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 2 | 2
Angina pectoris (Cardiac disorders) | 0 | 3 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 2
Conjunctival Haemorrhage (Eye disorders) | 12 | 21 | 2
Punctate Keratitis (Eye disorders) | 5 | 1 | 0
Eye Pain (Eye disorders) | 5 | 1 | 1
Vitreous Floaters (Eye disorders) | 3 | 2 | 0
Cataract (Eye disorders) | 4 | 3 | 1
Retinal Haemorrhage (Eye disorders) | 3 | 3 | 2
Posterior Capsule Opacification (Eye disorders) | 3 | 0 | 0
Visual Acuity Reduced (Eye disorders) | 3 | 3 | 0
Conjunctival Hyperaemia (Eye disorders) | 3 | 7 | 3
Vitreous Haemorrhage (Eye disorders) | 2 | 3 | 0
Vitreous Detachment (Eye disorders) | 2 | 1 | 2
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 3 | 2
Nausea (Gastrointestinal disorders) | 0 | 3 | 3
Sinusitis (Infections and infestations) | 4 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 3 | 5 | 2
Ear Infection (Infections and infestations) | 1 | 2 | 2
Pneumonia (Infections and infestations) | 1 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Syncope (Nervous system disorders) | 3 | 1 | 2
Cerebrovascular Accident (Nervous system disorders) | 1 | 3 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 2
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 2 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.